CLINICAL TRIAL: NCT04830033
Title: A Randomised Controlled Trial of the English National Opera Breathe Programme Compared With Usual Care in People Recovering From COVID-19
Brief Title: ENO Breathe vs Usual Care in COVID-19 Recovery
Acronym: SHIELD ENO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHIELD COVID - ENO sub-study 2
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Recovery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking of participants not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENO Breathe group (Experimental): Participation in the online ENO Breathe programme for 6 weeks.
  Interventions: Other: ENO Breathe group
- Usual Care Group (No Intervention): Participants continue with usual care.

INTERVENTIONS:
Other: ENO Breathe group — Six weekly group online workshop sessions, led by an ENO vocal specialist. Workshops will encourage participants to take part in exercises and activities especially designed to support breathing control, providing tools for self-management of breath and anxiety. They will also have access to bespoke online digital resources, designed to support participants between sessions. These will include exercises, song sheets and audio and video materials, especially recorded by the ENO for participants on the programme.
  Arms: ENO Breathe group

SUMMARY:
A randomised clinical trial to assess the impact of an online singing, breathing and wellbeing programme (ENO Breathe) developed specifically for people recovering from COVID-19.

DETAILED DESCRIPTION:
BACKGROUND:

ENO Breathe is a breathing and wellbeing programme developed specifically for people recovering from COVID-19, who are still suffering from breathlessness and associated anxiety. Delivered by ENO in collaboration with Imperial College Healthcare teams entirely online, the programme focuses on breathing re-training through singing. Initial evaluation of the project suggested health improvements related to participation, however, a properly conducted efficacy study is needed.

DESIGN: An assessor blind, parallel group, randomised controlled trial, to assess the effects of ENO Breathe compared to usual care on health status. The study will also evaluate the impact on respiratory symptoms, anxiety, depression, and breathlessness perception to investigate the mechanisms involved.

RESEARCH QUESION AND OUTCOME MEASURES:

The primary outcome will be change in health status, assessed using the RAND-36 tool (RAND SF-36), comparing ENO Breathe and Usual Care arms.

Additional endpoints will be: the COPD assessment test score (CAT), 0-100 Visual Analogue Scales (VAS) for breathlessness (at rest, walking around the house, climbing stairs, and running), Dyspnoea-12, anxiety (GAD-7), and depression (PHQ-9).

Assessments: The outcomes outlined above will be recorded at baseline prior to randomisation, and then repeated after 6 weeks.

POPULATION: Adult patients recovering from COVID-19 will be recruited from specialist COVID-19 clinics, where participants will have been fully assessed and investigated by referring healthcare professionals. Participants in the active arm will attend once weekly ENO online workshop sessions for 6 weeks, and have access to bespoke online digital resources, designed to support participants between sessions. The comparison arm will receive usual care. Randomization will be 1:1.

SAMPLE SIZE Sample size: Based on pilot data in people with COPD, where the standard deviation (SD) for change in SF-36 was 15 points, to identify a clinically relevant 10 point difference in SF-36 responses at a 0.05 level of significance with a 90% power would require 48 patients in each treatment arm. Allowing for 20% dropout, we will therefore recruit 120 patients.

Primary analysis will be on an intention to treat basis. Change in parameters will be assessed comparing ENO Breathe and Usual Care, using Generalised Linear Models to estimate treatment effects. In order to better understand changes in the RAND-36 "anchor measure", the investigator will relate this to changes in measures of anxiety, depression, breathlessness, and other respiratory symptoms.

An additional responder analysis will compare the proportion in each treatment arm achieving a clinically important (10%) improvement in RAND-36 scores.

Update 21 JUNE 2021

To calculate the sample size, pilot data from a singing-based intervention in COPD, (considered the most relevant data available at study inception) was used, as outlined above, where the researchers aimed to recruit 120 patients. Data subsequently became available from ENO Breathe participants that rook part in the program prior to the research study, in which the SD was 8 for change in SF-36 scores. We have also decided using an MCID of 5 for the SF-36 is more appropriate, as this is not specific to a particular medical condition. As such, a total sample of 108 participants is required, using 1 to 1 study arm allocation. Allowing for 30% dropout, which is more appropriate, 158 participants will be recruited. Additionally, as a higher than expected number of participants were considered, study withdrawals due to be unable to attend the session times they were allocated, or despite meeting inclusion criteria, 1-to-1 meeting with the session leaders highlighted issues related excessive fatigue precipitated by exertion, so were not deemed appropriate at that point in time. As such, the researchers will also conduct a modified intention to treat analysis including all participants who were randomised and were deemed appropriate to participate following their 1-to-1. This consideration had not been included in the original exclusion criteria, due to limited awareness of its relevance at that time. These changes have been made, and here documented, before any baseline data has been sent to the analysis team, and before any follow up data has been collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults recovering from COVID-19 with ongoing breathlessness and/or anxiety.
* Referred from a specialist COVID-19 clinics aligned with the project, after appropriate clinical evaluation and investigation
* Internet access with appropriate device (e.g. computer or tablet)

Exclusion Criteria:

- Unable to participate due to comorbidity (e.g. life limiting illness, cognitive impairment)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in RAND-36 (RAND SF-36) | At baseline, then repeated after 6 weeks.
  A well-established, supervised, self-completion health status questionnaire. This consists of eight sections for which a score of 0 to 100 is created, with 0 being maximum disability and 100 equivalent to no disability.

SECONDARY OUTCOMES:
Changes in COPD assessment test (CAT) | At baseline, then repeated after 6 weeks.
  A respiratory disease health status measure that has been validated in people recovering from COVID-19. This includes 8 items, scored 0-5 with a possible score from 0 (best) to 40 (worst).
Changes in Generalised Anxiety Disorder Assessment (GAD-7) | At baseline, then repeated after 6 weeks.
  Self-administered questionnaire to assess for symptoms, and severity, of anxiety. Includes seven questions scored from 0 to 3, giving a total score out of 21. Lower scores indicate less symptoms of anxiety.
Changes in Patient Health Questionnaire 9 (PHQ-9) | At baseline, then repeated after 6 weeks.
  Self-administered questionnaire to assess for symptoms, and severity, of depression. Includes nine questions scored from 0 to 3, giving a total score out of 27. Lower scores indicate less symptoms of depression.
Changes in Dyspnoea-12 questionnaire | At baseline, then repeated after 6 weeks.
  Assessment of dyspnoea. Includes 12 descriptors scored from 0 to 3, giving a total score of 36. Lower scores indicate less severe dyspnoea.
Changes in Visual Analogue Scale ratings of breathlessness | At baseline, then repeated after 6 weeks.
  Four Visual Analogue Scales, scored from 0 to 100, for participants to rate their breathlessness while i) at rest, ii) walking around the house, iii) climbing stairs, iv) running. Higher scores indicate more severe dyspnoea (breathlessness).
Changes in SF-6D (Short-Form Six-Dimension) scores | At baseline, then repeated after 6 weeks.
  The SF-6D uses data from the RAND SF-36 to generate a continuous index for health that can be used to create a quality-of-life score for cost utility analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hopkinson, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on reasonable request.
Supporting Information: Study Protocol
Time Frame: The data will be available from the date of publication of the main study, and will remain available for at least 2 years.
Access Criteria: Data will be shared on reasonable request.

REFERENCES:
- [Derived] Philip KEJ, Owles H, McVey S, Pagnuco T, Bruce K, Brunjes H, Banya W, Mollica J, Lound A, Zumpe S, Abrahams AM, Padmanaban V, Hardy TH, Lewis A, Lalvani A, Elkin S, Hopkinson NS. An online breathing and wellbeing programme (ENO Breathe) for people with persistent symptoms following COVID-19: a parallel-group, single-blind, randomised controlled trial. Lancet Respir Med. 2022 Sep;10(9):851-862. doi: 10.1016/S2213-2600(22)00125-4. Epub 2022 Apr 27. PMID 35489367